CLINICAL TRIAL: NCT07292753
Title: Role of Vitamin D Supplementation Versus Desmopressin Versus Their Combination in the Treatment of Primary Monosymptomatic Nocturnal Enuresis in Children With Vitamin D Deficiency: A Randomized Clinical Trial
Brief Title: Vitamin D Versus Desmopressin Versus Combination Therapy in Children With Primary Monosymptomatic Nocturnal Enuresis and Vitamin D Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ibrahim Magdy Ibrahim Mohammed, Resident of Urology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU_MS402_2025
Record Dates: First submitted 2025-12-06; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Nocturnal Enuresis; Vitamin D Deficiency
Keywords: Primary monosymptomatic nocturnal enuresis; Bedwetting; Pediatric nocturnal enuresis; Desmopressin; Vitamin D supplementation; Vitamin D deficiency; Pediatric urology; Children 6-12 years; Randomized clinical trial
MeSH Terms: conditions — Nocturnal Enuresis; Vitamin D Deficiency | interventions — Vitamin D; Deamino Arginine Vasopressin

STUDY DESIGN:
Intervention Model Description: Three-arm parallel-group randomized trial comparing vitamin D alone, desmopressin alone, and their combination in children with primary monosymptomatic nocturnal enuresis and vitamin D deficiency.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vitamin D Monotherapy (Experimental): Participants receive vitamin D supplementation at a dose of 2000 IU orally once daily for 6-12 weeks, followed by a maintenance dose of 600 IU orally once daily for the remainder of the 6-month treatment period.
  Interventions: Drug: Vitamin D
- Desmopressin Monotherapy (Active Comparator): Participants receive desmopressin 0.2 mg orally once daily at bedtime for the full 6-month treatment period. Dose adjustments follow standard pediatric nocturnal enuresis guidance if needed.
  Interventions: Drug: Desmopressin
- Combination Therapy (Vitamin D + Desmopressin) (Experimental): Participants receive vitamin D supplementation (2000 IU orally once daily for 6-12 weeks, then 600 IU daily) combined with desmopressin 0.2 mg orally once daily at bedtime for a total of 6 months.
  Interventions: Drug: Vitamin D; Drug: Desmopressin

INTERVENTIONS:
Drug: Vitamin D — Oral vitamin D supplementation used to correct vitamin D deficiency in children with primary monosymptomatic nocturnal enuresis.
  Arms: Combination Therapy (Vitamin D + Desmopressin); Vitamin D Monotherapy
Drug: Desmopressin — Oral desmopressin used as antidiuretic therapy for primary monosymptomatic nocturnal enuresis in children.
  Arms: Combination Therapy (Vitamin D + Desmopressin); Desmopressin Monotherapy

SUMMARY:
This randomized clinical trial evaluated three treatment approaches for children aged 6 to 12 years who had primary monosymptomatic nocturnal enuresis (night-time bedwetting) and confirmed vitamin D deficiency. Bedwetting is common in school-aged children and can affect self-esteem, social interactions, and school performance. Although desmopressin is widely used, some children do not respond adequately. Previous studies suggested that low vitamin D levels might contribute to bedwetting, raising the possibility that vitamin D supplementation could help.

In this study, eligible children were randomly assigned to one of three groups:

1. vitamin D supplementation alone,
2. desmopressin alone, or
3. a combination of vitamin D and desmopressin.

All participants were followed for up to six months. The primary aim was to compare the improvement in the number of wet nights per week among the three groups. Secondary assessments included treatment tolerability, changes in vitamin D levels, changes in serum sodium, and any treatment-related side effects.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 6 to 12 years
* Primary monosymptomatic nocturnal enuresis
* At least 2 episodes of night-time bedwetting per week for ≥3 consecutive months
* Serum 25-hydroxyvitamin D level <20 ng/mL
* Normal kidney function
* Normal serum sodium level
* Absence of daytime lower urinary tract symptoms (urgency, frequency, dysuria)
* Informed consent from parent or guardian and assent from the child when appropriate

Exclusion Criteria:

* Non-monosymptomatic nocturnal enuresis (daytime storage or voiding symptoms)
* Congenital urinary tract anomalies (e.g., meatal stenosis, hypospadias, epispadias)
* Urinary tract infection until culture becomes negative
* Neurological abnormalities, including suspected neurogenic bladder
* Endocrine diseases such as diabetes mellitus or hyperthyroidism
* Congestive heart failure or significant cardiac disease
* Prior or current use of vitamin D supplementation
* Serum sodium below normal range
* Chronic systemic illness
* Any condition judged by investigators to interfere with study participation

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Change in number of wet nights per week at 3 months | Baseline and 3 months after initiation of therapy
  Mean change in the number of nocturnal enuresis (bedwetting) episodes per week from baseline to 3 months after starting treatment, comparing the three groups (vitamin D alone, desmopressin alone, and combination therapy).

SECONDARY OUTCOMES:
Change in number of wet nights per week at 6 months | Baseline and 6 months after initiation of therapy
  Mean change in the number of nocturnal enuresis episodes per week from baseline to 6 months after starting treatment, comparing the three treatment groups.
Proportion of patients with complete response at 3 and 6 months | 3 months and 6 months after initiation of therapy
  Percentage of participants who achieve complete response, defined as 0 wet nights per week compared with baseline.
Proportion of patients with partial response at 3 and 6 months | 3 months and 6 months after initiation of therapy
  Percentage of participants who achieve partial response, defined as a ≥50% reduction in the number of wet nights per week compared with baseline.
Change in serum sodium level | Baseline, 1 week, 1 month, 3 months, and 6 months after initiation of desmopressin therapy
  Mean change in serum sodium concentration from baseline to follow-up visits and proportion of patients developing hyponatremia in each treatment group.
Change in serum 25-hydroxyvitamin D level | Baseline, 1 month, 3 months, and 6 months after initiation of therapy
  Mean change in serum 25(OH) vitamin D concentration from baseline to follow-up visits in each treatment group.
Incidence of hyponatremia | Baseline to 6 months after initiation of therapy
  Number and percentage of participants who develop hyponatremia (serum sodium below normal range) during the study period.
Incidence of headache | Baseline to 6 months
  Number and percentage of participants reporting headache that begins after treatment initiation and is considered treatment-related.
Incidence of gastrointestinal symptoms | Baseline to 6 months
  Number and percentage of participants reporting nausea, abdominal discomfort, or other gastrointestinal symptoms considered related to treatment.
Incidence of polyuria | Baseline to 6 months
  Number and percentage of participants who develop polyuria or clinically significant increase in urine output associated with therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the study results may be shared with qualified researchers upon reasonable request. Shared data will include variables necessary to confirm the primary and secondary outcome analyses. No information that could identify participants will be provided.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available beginning 6 months after publication of the study results and will remain available for 3 years thereafter.
Access Criteria: Researchers must submit a methodologically sound proposal outlining the intended use of the data. Access will be granted after review and approval by the study's principal investigator and the ethics committee. A data use agreement will be required before data are released.